CLINICAL TRIAL: NCT01797094
Title: BOTOX® in the Treatment of Upper Facial Lines in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191622-122
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-01

CONDITIONS: Upper Facial Rhytides; Crow's Feet Lines; Glabellar Lines; Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin Type A (44U) (Experimental): 44 units (U) botulinum toxin Type A (total dose) per treatment. 24 U injected into bilateral Crow's Feet Line areas and 20 U injected into Frown Line area on Day 1. Based on retreatment criteria participants were eligible for up to 5 treatment cycles.
  Interventions: Biological: botulinum toxin Type A (44U)
- Botulinum toxin Type A (32U) (Experimental): 32 units (U) botulinum toxin Type A (total dose) per treatment. 12 U injected into bilateral Crow's Feet Line areas and 20 U injected into Frown Line area on Day 1. Based on retreatment criteria participants were eligible for up to 5 treatment cycles.
  Interventions: Biological: botulinum toxin Type A (32U)

INTERVENTIONS:
Biological: botulinum toxin Type A (44U) — 44 units botulinum toxin Type A (total dose) per treatment. 24 U injected into bilateral Crow's Feet Line areas and 20 U injected into Frown Line area.
  Other Names: BOTOX®
  Arms: Botulinum toxin Type A (44U)
Biological: botulinum toxin Type A (32U) — 32 units botulinum toxin Type A (total dose) per treatment. 12 U injected into bilateral Crow's Feet Line areas and 20 U injected into Frown Line area.
  Other Names: BOTOX®
  Arms: Botulinum toxin Type A (32U)

SUMMARY:
This study will evaluate the safety and efficacy of BOTOX® (botulinum toxin Type A) for the treatment of upper facial lines (Crow's Feet Lines and Frown Lines).

ELIGIBILITY:
Inclusion Criteria:

-Moderate to severe Crow's Feet Lines and Frown Lines

Exclusion Criteria:

* Current or previous botulinum toxin treatment of any serotype
* Diagnosis of Myasthenia gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis
* Facial laser or light treatment for cosmetic purposes, microdermabrasion, superficial peels, or topical retinoid therapy or hormone cream within 3 months
* Laser treatment or phototherapy of the face for medical purposes, blepharoplasty, brow-lift or related procedure, periorbital permanent make-up, or oral retinoid therapy within one year
* Medium-depth or deep facial peels within 5 years
* Prior facial cosmetic surgery (e.g., prior periorbital surgery, facial lift, periorbital treatment with fillers, implantation or transplantation)

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Botulinum Toxin Type A (44U): 44 units (U) botulinum toxin Type A (total dose) per treatment. 24U injected into bilateral Crow's Feet Line areas and 20U injected into Frown Line area on Day 1. Based on retreatment criteria participants were eligible for up to 5 treatment cycles.
- Botulinum Toxin Type A (32U): 32 units (U) botulinum toxin Type A (total dose) per treatment. 12U injected into bilateral Crow's Feet Line areas and 20U injected into Frown Line area on Day 1. Based on retreatment criteria participants were eligible for up to 5 treatment cycles.
Period: Overall Study
Arm/Group | Botulinum Toxin Type A (44U) | Botulinum Toxin Type A (32U)
Started | 48 | 53
Completed | 42 | 51
Not Completed | 6 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Personal Reasons | 4 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Other Miscellaneous Reasons | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A (44U) | Botulinum Toxin Type A (32U) | Total
Number analyzed (Participants) | 48 | 53 | 101
Age, Customized [Number; unit: participants]
  ≤ 50 years | 29 | 40 | 69
  > 50 years | 19 | 13 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 48 | 93
  Male | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving None or Mild on the Investigator's Assessment of the Severity of Crow's Feet Lines (CFL) at Maximum Smile Using the Facial Wrinkle Scale-Asian (FWS-A)
Description: The Investigator assessed the severity of the participant's Crow's Feet lines at maximum smile using the 4-point Facial Wrinkle Scale where 0=none, 1=mild, 2=moderate or 3=severe. The percentage of participants with a score of none or mild at Day 30 is reported.
Time Frame: Day 30
Population: Intent-to-treat population included all enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Botulinum Toxin Type A (44U) | Botulinum Toxin Type A (32U)
Number analyzed (Participants) | 48 | 53
percentage of participants | 89.6 | 84.9

2. Secondary Outcome: Percentage of Participants Much Improved or Very Much Improved in the Subject's Assessment of Appearance of CFL as Measured by the Global Assessment of Change in Crow's Feet Lines (SGA-CFL)
Description: Participants rated the change in their Crow's Feet Lines using the SGA-CFL 7-point scale where 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse or 7=very much worse at Day 30. The percentage of participants who reported Much Improved or Very Much Improved at Day 30 is reported.
Time Frame: Day 30
Population: Intent-to-treat population included all enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Botulinum Toxin Type A (44U) | Botulinum Toxin Type A (32U)
Number analyzed (Participants) | 48 | 53
percentage of participants | 87.6 | 77.4

3. Secondary Outcome: Percentage of Participants With a ≥2-Point Improvement From Baseline for Facial Line Outcomes Questionnaire (FLO-11) Item 2 at Day 30
Description: The FLO-11 questionnaire is comprised of 11 items that assess the subject's perceptions about specific aspects of their facial lines for the previous 7 days. Each question was scored on an 11-point scale (0=not at all, 5=somewhat, 10=very much). FLO-11 responders were defined as the percentage of participants with a ≥2-point improvement from Baseline in FLO-11 Item 2 : "When I look in the mirror, my facial lines make me look older than I want to look" score.
Time Frame: Baseline, Day 30
Population: Intent-to-treat population included all enrolled participants. Only participants with FLO-11 Item 2 scores ≥2 at Baseline are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Botulinum Toxin Type A (44U) | Botulinum Toxin Type A (32U)
Number analyzed (Participants) | 46 | 50
percentage of participants | 84.8 | 88.0

4. Secondary Outcome: Percentage of Participants With a ≥2-point Improvement From Baseline for Facial Line Outcomes Questionnaire (FLO-11) Item 5 at Day 30
Description: The FLO-11 questionnaire is comprised of 11 items that assess the subject's perceptions about specific aspects of their facial lines for the previous 7 days. Each question was scored using an 11-point scale (0=not at all, 5=somewhat, 10=very much). FLO-11 responders were defined as the percentage of participants with a ≥2-point improvement from Baseline in FLO-11 Score Item 5: "My facial lines make me look less attractive than I want to look" score.
Time Frame: Baseline, Day 30
Population: Intent-to-treat population included all enrolled participants. Only participants with FLO-11 Item 5 scores ≥2 at Baseline are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Botulinum Toxin Type A (44U) | Botulinum Toxin Type A (32U)
Number analyzed (Participants) | 46 | 51
percentage of participants | 73.9 | 72.5

5. Secondary Outcome: Percentage of Participants With a ≥3-Point Improvement From Baseline for Facial Line Outcomes Questionnaire (FLO-11) Item 8 at Day 30
Description: The FLO-11 questionnaire is comprised of 11 items that assess the subject's perceptions about specific aspects of their facial lines for the previous 7 days. Each question was scored on an 11-point scale (0=not at all, 5=somewhat, 10=very much) FLO-11 responders were defined as the percentage of participants with a ≥3-point improvement from Baseline in FLO-11 Item 8: "My facial lines make me look tired" score.
Time Frame: Baseline, Day 30
Population: Intent-to-treat population included all enrolled participants. Only participants with FLO-11 Item 8 scores ≥ 3 at Baseline were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Botulinum Toxin Type A (44U) | Botulinum Toxin Type A (32U)
Number analyzed (Participants) | 43 | 49
percentage of participants | 86.0 | 69.4

6. Secondary Outcome: Percentage of Participants Who Rate Themselves in a Younger Self-Perception of Age Category Than at Baseline
Description: Participants were considered to judge themselves as looking younger if the category change was from "look my current age" at Baseline to "look younger" at Day 30 or from "look older" at Baseline to "look my current age/younger" at Day 30.
Time Frame: Baseline, Day 30
Population: Intent-to-treat population included all enrolled participants. Only those participants who rated themselves as looking their current age or older at Baseline were included in the analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Botulinum Toxin Type A (44U) | Botulinum Toxin Type A (32U)
Number analyzed (Participants) | 46 | 51
percentage of participants | 54.3 | 56.9

7. Secondary Outcome: Percentage of Participants Mostly or Very Satisfied With Their Crow's Feet Lines on the Facial Line Satisfaction Questionnaire
Description: Participants assessed their overall satisfaction at the present moment using a 5-point scale where -2=very dissatisfied, -1=mostly dissatisfied, 0=neither dissatisfied nor satisfied, 1=mostly satisfied and 2=very satisfied. The percentage of participants mostly or very satisfied is reported.
Time Frame: Day 30
Population: Intent-to-treat population included all enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Botulinum Toxin Type A (44U) | Botulinum Toxin Type A (32U)
Number analyzed (Participants) | 48 | 53
percentage of participants | 81.3 | 81.1

ADVERSE EVENTS:
Description: The Safety Population, all enrolled participants who received study drug, was used to determine the number of participants at risk for Serious Adverse Events and Adverse Events.
Arm/Group | Botulinum Toxin Type A (44U) | Botulinum Toxin Type A (32U)
Serious Adverse Events (participants affected / at risk) | 1/47 | 4/53
Other Adverse Events (participants affected / at risk) | 20/47 | 22/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Botulinum Toxin Type A (44U) (N=47) | Botulinum Toxin Type A (32U) (N=53)
Hepatitis A (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bartholin's cyst (Reproductive system and breast disorders) | 0/44 | 1/48 — Female population only.
Benign female reproductive tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/44 | 1/48 — Female population only.
Peritonitis (Infections and infestations) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (44U) (N=47) | Botulinum Toxin Type A (32U) (N=53)
Injection site haemorrhage (General disorders) | 9 | 6
Nasopharyngitis (Infections and infestations) | 5 | 6
Eyelid ptosis (Eye disorders) | 4 | 2
Eczema (Skin and subcutaneous tissue disorders) | 2 | 5
Pharyngitis (Infections and infestations) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.